CLINICAL TRIAL: NCT04321538
Title: Evaluation of the GoCheck Kids Mobile Vision Screening Application and the Welch Allyn Spot Vision Screener
Brief Title: Gocheck Kids vs. Welch Allyn Spot Vision Screener
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000026666
Record Dates: First submitted 2020-03-24; First posted 2020-03-25 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Amblyopia
Keywords: GoCheck Kids; Welch Allyn Spot Vision Screener; Vision Screening; Photoscreening
MeSH Terms: conditions — Amblyopia | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Failed Vision Screen Cohort: This cohort represents the entire group of study participants- children who were referred to Yale New Haven Hospital and Yale Medicine for a failed vision screen by either their primary care provider or their school.
  Interventions: Device: Gocheck Kids; Device: Welch Allyn Spot Vision Screener; Diagnostic Test: Physical Exam

INTERVENTIONS:
Device: Gocheck Kids — GoCheck Kids is a photoscreening device. It takes a special picture of the eyes that allows for detection of refractive error and eye misalignment.
Device: Welch Allyn Spot Vision Screener — The Welch Allyn Spot Vision Screener is a photoscreening device. It takes a special picture of the eyes that allows for the detection of refractive error and eye misalignment.
Diagnostic Test: Physical Exam — Retinoscopy and an oculomotor testing will constitute the physical examination.

SUMMARY:
The investigators are conducting a prospective evaluation of the ability of two vision photoscreening devices (GoCheck Kids and the Welch Allyn Spot Vision Screener) to detect risk factors for amblyopia. Photoscreeners function similar to having a picture taken with a camera. Amblyopia is decreased vision in one or both eyes due to decreased vision development in the brain resulting from decreased visual stimulation. Children ages 1 year to less than 7 years of age referred to a pediatric ophthalmologist at Yale New Haven Health and Yale Medicine locations for a failed vision screen will be offered participation. The ability of each screening device to detect amblyopia risk factors will be compared with the results of a complete eye exam performed by the practitioner.

DETAILED DESCRIPTION:
The United States Preventive Services Task Force has recommended early screening in children in order to detect vision abnormalities that could result in amblyopia, a condition in which there is abnormal brain development when there is suboptimal vision in one or both eyes. Prior to the introduction of vision screening instruments, physicians would wait to screen children at age 3-4, when they are able to read letter or symbol charts. The introduction of vision screening instruments has provided a screening option for children as young as 6 months.

Photoscreening devices evaluate for amblyopia risk factors, including refractive error (need for glasses), or strabismus (eye misalignment). Since the advent of instrumental vision screening, improvements are continually being made to improve the quality and scope of vision screening devices. As more affordable and convenient instruments are developed to supplement the traditional letter charts used to screen children, there is a need for more prospective trials to test the efficacy of these instruments. Our study is designed to evaluate the latest model of GoCheck Kids iPhone vision screener with the widely-used Welch Allyn Spot Vision Screener. The GoCheck Kids smartphone application is paid for on a monthly basis and includes telephone rental rather than requiring that a device be purchased. This lower upfront cost option will allow for more primary care practices to participate with a decreased upfront financial burden.

Children ages 1 year to less than 7 years referred to a Yale New Haven Hospital and Yale Medicine pediatric ophthalmology practice for a failed vision screen will be prospectively recruited for participation at the time of their already scheduled appointment for a complete eye exam. Following informed consent, each participant will be screened using both the GoCheck Kids smartphone application and the Welch Allyn Spot Vision Screener. Screening for each of these devices involves a process akin to having a photograph taken. Obtaining consent and photo screenings will take less than 5 minutes. The complete eye exam, which will be performed in this referral group regardless of study participation, will include evaluation of the front and back of the eye, eye alignment, and determination of the refractive state by retinoscopy (check if glasses are needed by using a special type of light and handheld lenses). The ability of each screening device to detect amblyopia risk factors when they are present (sensitivity) will be determined by comparison with the detection of amblyopia risk factors during the complete eye exam, which is considered the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 1-<7 years.

Exclusion Criteria:

* Children with a history of ocular surgery and children with ocular conditions or behavior that preclude obtainment of the screening photo images or completion of a complete eye exam.
* Children with an obstructed visual axis.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 1-<7 years referred to a Yale New Haven Hospital and Yale Medicine associated pediatric ophthalmology practice for a failed vision screen.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Sensitivities for amblyopia risk factor detection | Up to 2 hours
  The sensitivity is the percentage of patients with amblyopia whose vision screen indicates they have an amblyopia risk factor. The sensitivity for the detection of amblyopia risk factors is determined individually for both the GoCheck Kids application and the Welch Allyn Spot Vision Screener by calculating the number of truly positive failed vision screens by the photoscreener (as determined by the gold standard physical exam including cycloplegic retinoscopy to look for refractive error and oculomotor exam to evaluate strabismus) and dividing by the sum of truly positive failed vision screens plus false-negative vision screens (the vision screener did not detect amblyopia risk factors when they were found to be present on the physical exam).

SECONDARY OUTCOMES:
Sensitivity for detection of refractive error | Up to 2 hours
  The refractive error will be determined using the gold standard physical exam technique of cycloplegic retinoscopy. The sensitivity for the detection of refractive error will be determined individually for both the GoCheck Kids application and the Welch Allyn Spot Vision Screener by calculating the number of truly positive failed vision screens for refractive error and dividing by the sum of truly positive failed vision screens for refractive error plus false-negative vision screens for refractive error.
Sensitivity for detection of strabismus | Up to 2 hours
  The presence of strabismus will be determined using an oculomolotor exam. The sensitivity for the detection of strabismus will be determined individually for both the GoCheck Kids application and the Welch Allyn Spot Vision Screener by calculating the number of truly positive failed vision screens for strabismus and dividing by the sum of truly positive failed vision screens for strabismus plus false-negative vision screens for strabismus.

CONTACTS AND LOCATIONS:
Overall Officials: Martha A Howard, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan on sharing protected health information with other researchers.

REFERENCES:
- [Background] US Preventive Services Task Force; Grossman DC, Curry SJ, Owens DK, Barry MJ, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW. Vision Screening in Children Aged 6 Months to 5 Years: US Preventive Services Task Force Recommendation Statement. JAMA. 2017 Sep 5;318(9):836-844. doi: 10.1001/jama.2017.11260. PMID 28873168